CLINICAL TRIAL: NCT02676648
Title: Randomized Trial of Web-Delivered Interventions for Blood Sugar Control for Individuals With Type 2 Diabetes
Brief Title: Web-Delivered Interventions for Blood Sugar Control for Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00102827
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Experimental: Condition 1 (Experimental): 1) core program; 2) breath meter; 3) text messages; 4) diet-appropriate food and cookbooks
  Interventions: Behavioral: Multicomponent online program; Behavioral: Breath meter; Behavioral: Text messages; Behavioral: Diet-appropriate foods and cookbooks
- Experimental: Condition 2 (Experimental): 1) core program
  Interventions: Behavioral: Multicomponent online program
- Experimental: Condition 3 (Experimental): 1) core program; 2) breath meter
  Interventions: Behavioral: Multicomponent online program; Behavioral: Breath meter
- Experimental: Condition 4 (Experimental): 1) core program; 2) text messages
  Interventions: Behavioral: Multicomponent online program; Behavioral: Text messages
- Experimental: Condition 5 (Experimental): 1) core program; 2) diet-appropriate food and cookbooks
  Interventions: Behavioral: Multicomponent online program; Behavioral: Diet-appropriate foods and cookbooks
- Experimental: Condition 6 (Experimental): 1) core program; 2) breath meter; 3) text messages
  Interventions: Behavioral: Multicomponent online program; Behavioral: Breath meter; Behavioral: Text messages
- Experimental: Condition 7 (Experimental): 1) core program; 2) breath meter; 3) diet-appropriate food and cookbooks
  Interventions: Behavioral: Multicomponent online program; Behavioral: Breath meter; Behavioral: Diet-appropriate foods and cookbooks
- Experimental: Condition 8 (Experimental): 1) core program; 3) text messages; 4) diet-appropriate food and cookbooks
  Interventions: Behavioral: Multicomponent online program; Behavioral: Text messages; Behavioral: Diet-appropriate foods and cookbooks

INTERVENTIONS:
Behavioral: Multicomponent online program — The core program includes information developed in earlier research with individuals with type 2 diabetes, now modified for online delivery: very low-carbohydrate diet taught with lectures on video, handouts, quizzes, and surveys. We also teach participants about the importance of physical activity and adequate sleep, in addition to psychological skills (positive affect, mindful eating) intending to help with intervention adherence.
Behavioral: Breath meter — We will send participants a breath meter to test ketones in their breath, to assess dietary adherence.
  Arms: Experimental: Condition 1; Experimental: Condition 3; Experimental: Condition 6; Experimental: Condition 7
Behavioral: Text messages — We will send participants text messages, to support intervention adherence.
  Arms: Experimental: Condition 1; Experimental: Condition 4; Experimental: Condition 6; Experimental: Condition 8
Behavioral: Diet-appropriate foods and cookbooks — We will send participants diet-appropriate foods and cookbooks, to support intervention adherence.
  Arms: Experimental: Condition 1; Experimental: Condition 5; Experimental: Condition 7; Experimental: Condition 8

SUMMARY:
The goal of the research is to optimize an online and mobile multicomponent 12-month diet and lifestyle intervention for improving the blood glucose control of individuals with type 2 diabetes.

DETAILED DESCRIPTION:
The research will identify the most promising intervention components. The following components will be tested: dietary adherence testing with a breath meter, text messages, and diet-appropriate foods and cookbooks. The primary goal is to optimize the intervention by examining the HbA1c results at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese
* English-speaking
* diagnosis of type 2 diabetes (HbA1c > 6.5%)
* regular access to the internet and text messages

Exclusion Criteria:

* taking diabetes medications other than metformin
* being pregnant or breastfeeding
* currently undergoing cancer treatments
* untreated serious mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 months
  Change in HbA1c from baseline to 12 months post baseline

SECONDARY OUTCOMES:
Body Weight Percent Lost | 12 months
  Change in body weight percentage from baseline to 12 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Laura Saslow, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saslow LR, Moskowitz JT, Mason AE, Daubenmier J, Liestenfeltz B, Missel AL, Bayandorian H, Aikens JE, Kim S, Hecht FM. Intervention Enhancement Strategies Among Adults With Type 2 Diabetes in a Very Low-Carbohydrate Web-Based Program: Evaluating the Impact With a Randomized Trial. JMIR Diabetes. 2020 Sep 9;5(3):e15835. doi: 10.2196/15835. PMID 32902391